CLINICAL TRIAL: NCT03440606
Title: Development and Evaluation of a Novel Mindful-Compassion Art Therapy (MCAT) Supervision for Self-Care and Collegial Support Among End-of-Life Care Professionals in Singapore
Brief Title: A Novel Mindful-Compassion Art Therapy (MCAT) Supervision
Acronym: MCAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanyang Technological University (Other)
Collaborators: HCA Hospice Care (Other)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Assistant Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-2015-04-021
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: End-of-life Care
Keywords: Randomized Wait-List Control Trial; Mindful-Compassion Art Therapy Supervision; End-of-Life Care; Self-Care

STUDY DESIGN:
Intervention Model Description: participants will be randomly assigned to either the intervention or waitlist control group. Those assigned to in the intervention group will attend 6 weekly Mindful-Compassion Art Therapy supervision led by a credentialed art therapist and an experienced mindfulness practitioner at the training facilities of HCA. Each session will last for 3 hours and each group will consists of 15 participants. Outcome assessments will be conducted at two-time-points: immediately after intervention [T2] and four weeks post intervention [T3]. Those assigned to the waitlist control group will receive no intervention until approximately three month later; equivalent intervention and assessment procedures will be administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCAT Supervision Group (Experimental): The 6-week 3-hour Mindful-Compassion Art Therapy (MCAT) supervision will include intervention elements of brief psycho-education, weekly mindfulness mediation that serve as a foundation to foster creative art making, reflective writing, group sharing and discussion.
  Interventions: Behavioral: Mindful-Compassion Art Therapy Supervision
- Waitlist Control Group (Experimental): Those assigned to the waitlist control group will not receive Mindful-Compassion Art Therapy (MCAT) supervision until approximately 1.5 month later; equivalent intervention and assessment procedures will be administered.
  Interventions: Behavioral: Mindful-Compassion Art Therapy Supervision

INTERVENTIONS:
Behavioral: Mindful-Compassion Art Therapy Supervision — Each "Mindful-Compassion Art Therapy Supervision" group will focus on 3 major areas that cultivate self-care, resilience and communal support. The specific structure include: (1) Self-care and Stress Management in Week 1 and 2 (i.e., concept of mindfulness and art, the symbol of the mandala and its use in self-care, mindfulness practice and art); (2) Sharing of Clinical Expertise and Experiences in Week 3 and 4 (i.e., Create mindful art about one meaningful and one challenging patient/client interaction with small group discussion); and (3) Understanding Grief and Meaning-Making in Week 5 and 6 (i.e., Create mindful art representing a clinical encounter of mortality, and meaning-making from reflection on grief).

SUMMARY:
Background: The need for empathy and the difficulties of coping with morality when caring for the dying and the bereaved pose great psychological and spiritual strains. End-of-Life (EoL) care professionals including doctors, nurses and social workers are particularly prone to burnout given the intense emotional and existential nature of their work. Supervision is one important way to provide adequate support that focuses on both professional and personal competencies in working with death and loss. Previous research has provided strong evidence that support the inclusion of art therapy within supervision for it had effectively reduced burnout and enhanced emotional regulation. Combining the practice of mindfulness in art-therapy based supervision has immense potential to create a dynamic platform for self-care and collegial support, of which could ultimately cultivate sustained resilience, compassion and growth among those immersed the fields of hospice and palliative care.

Methods/Design: A randomized wait-list control trial design. 60 EoL care professionals were randomly allocated into one of two groups: (i) Intervention group (MCAT Supervision), and (ii) Control group (MCAT Supervision will be provided after the intervention group completed all supervision sessions). Both quantitative and qualitative outcomes were assessed at baseline, immediately after intervention, and four weeks post intervention. Primary outcome measure included level of burnout. Secondary outcomes included death attitude and fear of death, emotional awareness and regulation, resilience, compassion, and overall quality of life. Qualitative data were analyzed using Framework method.

Discussion: The integration of art and mindfulness practice to process the needs of professional EoL caregivers for self-care is a scarcely explored area in the field of hospice and palliative care in Singapore and in the international context. This pilot study proposes to develop and test a novel Mindful-Compassion Art Therapy (MCAT) Supervision for professional EoL caregivers. The expected outcome would generate new knowledge contributing to advancements in both theories and practice in hospice and palliative care for Singapore and across the globe.

DETAILED DESCRIPTION:
Study Design

Building on the established protocol of Art-Therapy based supervision together with the additional elements of mindfulness practice, this study will adopt an randomized wait-list control trial design comprising of two groups: (i) Intervention group (MCAT Supervision), and (ii) Control group (MCAT Supervision will be provided after the intervention group completed all supervision sessions).

Study Site

Participants will be recruited from a community-based collaborating partner, Hospice Care Association (HCA), Singapore's largest home hospice care provider. Deputy Medical Director and Programme Director of HCA Star PALs, together with his appointed staffs will provide assistance in recruitment as well as tracking of participants, allowing for timely intervention and efficient data collection.

Participants

The sample will comprise of 60 frontline EoL caregivers including doctors, nurses, social workers and allied health professionals currently working in field of hospice and palliative care (N=60).

Allowing for an attrition rate of 15% at follow-up, a sample of 60 will provide 80% power to detect an effect size of 0.80 standard deviation units in the primary outcome measure of Maslach Burnout Inventory-General Survey between the intervention and control group at the (two-tailed test) 5% level of significance.

Recruitment, assessment, intervention, and follow up procedures

Upon informed consent and baseline assessment [T1] conducted via paper or electronic online questionnaires, participants will be randomly assigned to either the intervention or waitlist control group. Those assigned to in the intervention group will attend 6 weekly Mindful-Compassion Art Therapy supervision led by a credentialed art therapist and an experienced mindfulness practitioner at the training facilities of HCA. Each session will last for 3 hours and each group will consists of 15 participants. Outcome assessments will be conducted at two-time-points: immediately after intervention [T2] and four weeks post intervention [T3]. Those assigned to the waitlist control group will receive no intervention until approximately three month later; equivalent intervention and assessment procedures will be administered. The 6-week 3-hour MCAT supervision will include elements of brief psycho-education, weekly mindful mediation that serve as a foundation to foster art making, reflective writing, group sharing and discussion.

Between and within participants comparisons of quantitative outcomes will be conducted and the appropriate effect size estimates reported. The intervention group and control group will be compared on the main outcome (i.e. burnout) and secondary outcomes (i.e. fear and negative attitudes of death, emotional awareness and regulation, resilience, compassion, and overall quality life). T2 and T3 assessments will be compared with baseline assessment. The intervention and control groups will also be compared on demographic characteristics with baseline measures; if necessary, they variables will be controlled in the analyses. The SPSS statistical software package will be used to manage the data.

The Framework method of analysis will be used to analyze qualitative data. 28 Analyses will be both deductive (from pre-set aims and objectives) and inductive (arising from participants view). This method tends to be more structured than some other methods of qualitative analysis and the process more explicit and more informed by a priori questions. It is designed so that it can be more easily understood and assessed by people other than the analyst, such as funding bodies, policy makers and participants. Throughout the analytical process we will use strategies to maximize credibility, criticality, and authenticity. The QSR NVIVO software package will be used to manage the data.

ELIGIBILITY:
Inclusion Criteria:

* Frontline EoL caregivers including doctors, nurses, social workers and allied health professionals
* Currently working in field of hospice and palliative care
* Fluent in both written and verbal English
* Able to provide informed consent
* Not suffering from major mental health problems

Exclusion Criteria:

* Not fluent in both written and verbal English
* Unable to provide informed consent
* Suffering from major mental health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline 'Maslach Burnout Inventory- General Survey (MBI-GS)' at immediate after intervention [T2] and 4 weeks follow-up [T3]. | It will be assessed at baseline [T1], immediately after intervention [T2], and four weeks post intervention [T3].
  This tool measures changes in level of burnout.

SECONDARY OUTCOMES:
Change from Baseline 'Death Attitude Profile-Revised (DAP-R)' at immediate after intervention [T2] and 4 weeks follow-up [T3]. | It will be assessed at baseline [T1], immediately after intervention [T2], and four weeks post intervention [T3].
  This tool measures death attitudes and fear of death.
Change from Baseline 'Five Facet Mindfulness Questionnaire (FFMQ)' at immediate after intervention [T2] and 4 weeks follow-up [T3]. | It will be assessed at baseline [T1], immediately after intervention [T2], and four weeks post intervention [T3].
  This tool measures emotional awareness and regulation.
Change at Baseline 'Ego Resilience Scale-Revised (ER89-R)' at immediate after intervention [T2] and 4 weeks follow-up [T3]. | It will be assessed at baseline [T1], immediately after intervention [T2], and four weeks post intervention [T3].
  This tool measures resilience.
Change at Baseline 'Self-Compassion Scale Short-Form (SCS-SF)' at immediate after intervention [T2] and 4 weeks follow-up [T3]. | It will be assessed at baseline [T1], immediately after intervention [T2], and four weeks post intervention [T3].
  This tool measures compassion.
Change at Baseline 'World Health Organization Quality of Life Scale-8 (WHOQoL-8)' at immediate after intervention [T2] and 4 weeks follow-up [T3]. | It will be assessed at baseline [T1], immediately after intervention [T2], and four weeks post intervention [T3].
  This tool measures overall quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Hau Yan Ho, PhD, EdD, Principal Investigator — Nanyang Technological University
Locations (1):
- HCA Hospice Care, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Potash JS, Chan F, Ho AH, Wang XL, Cheng C. A Model for Art Therapy-Based Supervision for End-of-Life Care Workers in Hong Kong. Death Stud. 2015 Jan-Jun;39(1-5):44-51. doi: 10.1080/07481187.2013.859187. Epub 2014 Jun 23. PMID 24870589
- [Derived] Ho AHY, Tan-Ho G, Ngo TA, Ong G, Chong PH, Dignadice D, Potash J. A Novel Mindful-Compassion Art-Based Therapy for Reducing Burnout and Promoting Resilience Among Healthcare Workers: Findings From a Waitlist Randomized Control Trial. Front Psychol. 2021 Oct 21;12:744443. doi: 10.3389/fpsyg.2021.744443. eCollection 2021. PMID 34744918
- [Derived] Ho AHY, Tan-Ho G, Ngo TA, Ong G, Chong PH, Dignadice D, Potash J. A novel mindful-compassion art therapy (MCAT) for reducing burnout and promoting resilience for end-of-life care professionals: a waitlist RCT protocol. Trials. 2019 Jul 8;20(1):406. doi: 10.1186/s13063-019-3533-y. PMID 31287010